CLINICAL TRIAL: NCT03354702
Title: The Impact of Aerobic Physical Activity on Aspects of Impulsivity and Negative Affectivity in Pathological Gamblers
Brief Title: Physical Activity Pathological Gamblers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: physical and pathological gamb
Record Dates: First submitted 2017-09-11; First posted 2017-11-28 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group aerobic activity (experimental) (Experimental): Group aerobic exercise (experimental). Patients perform aerobic exercise per 30 minutes (moderate intensity: 70% to 85% of estimated maximum heart rate), more 10 minutes stretching, once a week monitored and once without monitoring and patients have medical appointment with psychiatrist and make psychotherapy sessions.
  Interventions: Other: Aerobic
- Group stretching (control) (Active Comparator): Group stretching (control). Patients perform stretching per 30 minutes, once a week monitored and once without monitoring and patients have medical appointment with psychiatrist and make psychotherapy sessions
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Aerobic — Aerobic exercise Patients performs 8 sessions of aerobic exercise (walking / running),with monitoring and 8 sessions without monitoring totaling 16 sessions and patients have medical appointment with psychiatrist and make psychotherapy sessions.
  Arms: Group aerobic activity (experimental)
Other: Stretching — Stretching Patients performs 8 sessions of stretching, with monitoring and 8 sessions without monitoring totaling 16 sessions and patients have medical appointment with psychiatrist and make psychotherapy sessions.
  Arms: Group stretching (control)

SUMMARY:
Gambling Disorder (GD) is defined as the recurrent and persistent act of betting which leads to clinical impairments,. The latest edition of the Diagnostic and Statistical Manual of Mental Disorders (5th edition) conceptualizes GD as a behavioral addiction due to the similarities between GD and substance addictions in clinical presentation, association with personality factors, genetic transmission and treatment options. Previous studies found potential benefits of physical activity in treatment of addictions in general and GD in particular, such as reducing desire to play, betting and depressive and anxious symptoms.

DETAILED DESCRIPTION:
Detailed Description: The purpose of this study is to investigate the effects of regular physical activity controlled and supervised in the treatment of gambling disorder with focus on gambling severity, psychiatric comorbidity and impulsiveness. Patients will undergo physical activity either running (experimental) or stretching (control) groups,. Physical activity sessions will be lead by a physical educator., Both groups will receive treatment for psychiatric comorbidities and cognitive behavioral psychoeducation.

ELIGIBILITY:
Inclusion criteria:

* Five or more diagnostic criteria for pathological gambling specified in the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV-TR - APA, 2000);
* At least four years of formal education;
* Able to perform physical activity;
* Non-pregnant.

Exclusion criteria:

* Clinical pathology that demands urgent care such as hospitalization in another service;
* Any cardiorespiratory, musculoskeletal, or clinical condition that could prevent the practice of aerobic activity, established in clinical evaluation prior to randomization;
* Psychotic disorder that may undermine validity of responses to the self-report scales administered;
* Condition which affects the central nervous system and seriously impairs cognitive functions, as a disorder oligophrenia;
* Diagnosis of moderate to severe depression that compromises engagement in physical activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Gambling Follow-up scale (GFS) | Eight weeks
  This questionnaire is meant to assess gambling severity and it investigates financial issues, family relationships, emotional distress, and satisfaction with leisure, in addition to gambling behavior.
International Neuropsychiatric Interview | Eight weeks
  The MINI is a brief psychiatric interview that has strong psychometric properties including reliable diagnoses as compared to the Composite International Diagnostic Interview and the Structured Clinical Interview for the DSMpsychiatric disorder in axis I of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) of American Psychiatric Association in 1994. International Neuropsychiatric Interview takes approximately 15 minutes.

SECONDARY OUTCOMES:
Gambling Symptom Assessment Scale (GSA-S). | Eight weeks
  The G-SAS is a 12-item instrument which was designed to evaluate gambling symptoms. Each item is scored on a 5-point Likert scale from 0 'none' or 'complete' to 4 'extreme' or 'no control'. Scores range from 0 to 48 with four severity categories: mild (8-20), moderate (21-30), severe (31-40), and extreme (41-48).
Barratt Impulsiveness Scale (BIS-11) | Eight weeks
  It is a self-report scale consisting of 30 questions that provides a total score (minimum of 30 and maximum of 120) resulting from the sum of three sub-factors, namely: lack of attention, that is, cognitive impulsivity (i.e., decisions made in haste), motor impulsivity (i.e., acts without thinking) and non-planning (i.e., behaviors performed without future perspective).
GoStop Impulsivity Paradigm. | Eight weeks
  GoStop Impulsivity Paradigm evaluates the capacity of inhibitory control. GoStop Impulsivity Paradigm is a "stop task" designed to measure response inhibition. The primary response of interest here is the failure to inhibit responding when a "go" cue is unexpectedly accompanied by a "stop" cue.
Delay DiscountingTask (DDT). | Eight weeks
  In the Delay Discount Test (DDT) the subject is faced with a hypothetical choice, for example receiving US$ 1,000.00 in 6 hours, or US$ 999.00 now. The value of the present reward is presented in descending order until the subject chooses to wait for the delayed reward. The value immediately prior to this change is called the point of indifference.
The Rey-Osterrieth Complex Figure Test | Eight weeks
  The Rey-Osterrieth Complex Figure Test assesses visuospatial organization and planning abilities. The subject has to copy a complex geometric figure. A score is calculated for the drawing taking into account number of details, reproduction strategy, and drawing organization.

CONTACTS AND LOCATIONS:
Overall Officials: HERMANO TAVARES, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital da Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil